CLINICAL TRIAL: NCT02573259
Title: A PHASE 1, OPEN-LABEL, DOSE ESCALATION AND EXPANSION STUDY OF PF-06801591 IN PATIENTS WITH LOCALLY ADVANCED OR METASTATIC MELANOMA, SQUAMOUS CELL HEAD AND NECK CANCER, OVARIAN CANCER, SARCOMA, NON-SMALL CELL LUNG CANCER, UROTHELIAL CARCINOMA OR OTHER SOLID TUMORS.
Brief Title: A Dose Escalation Study Of PF-06801591 In Melanoma, Head And Neck Cancer (SCCHN), Ovarian, Sarcoma, Non-Small Cell Lung Cancer, Urothelial Carcinoma or Other Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: B8011001; 2016-003314-27 (EudraCT Number)
Record Dates: First submitted 2015-10-06; First posted 2015-10-09 (Estimated); Results first posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-10

CONDITIONS: Part 1; MELANOMA; SCCHN; OVCA; SARCOMA; OTHER SOLID TUMORS; Part 1 and 2; NSCLC; UROTHELIAL CARCINOMA
Keywords: efficacy; safety; pharmacokinetics; pharmacodynamics; open label; dose response; multiple ascending dose; immunogenicity; recommended phase 2 dose; subcutaneous
MeSH Terms: conditions — Melanoma; Sarcoma; Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 PF-06801591 (Experimental): 0.5 mg/kg IV every 21 days (Part 1)
  Interventions: Drug: PF-06801591
- Arm 2 PF-06801591 (Experimental): 1.0 mg/kg IV every 21 days (Part 1)
  Interventions: Drug: PF-06801591
- Arm 3 PF-06801591 (Experimental): 3.0 mg/kg IV every 21 days (Part 1)
  Interventions: Drug: PF-06801591
- Arm 4 PF-06801591 (Experimental): 10 mg/kg IV every 21 days (Part 1)
  Interventions: Drug: PF-06801591
- Arm 5 PF-06801591 (Experimental): 300 mg SC every 28 days (Part 1 and 2)
  Interventions: Drug: PF-06801591

INTERVENTIONS:
Drug: PF-06801591 — IV every 21 days (Part 1)
  Arms: Arm 1 PF-06801591; Arm 2 PF-06801591; Arm 3 PF-06801591; Arm 4 PF-06801591
Drug: PF-06801591 — 300 mg SC every 28 days (Part 1 and 2)
  Arms: Arm 5 PF-06801591

SUMMARY:
Protocol B8011001 is a Phase 1, open-label, multi-center, multiple-dose, dose escalation and expansion, safety, pharmacokinetics (PK), and pharmacodynamics (PD) study of PF-06801591 in previously treated adult patients with locally advanced or metastatic melanoma, SCCHN, ovarian carcinoma, sarcoma, NSCLC, urothelial carcinoma or other solid tumors. This is a 2 Part study whereby the safety and tolerability of increasing dose levels of intravenous (IV) or subcutaneous (SC) PF-06801591 was assessed in Part 1. Part 2 expansion is designed to further evaluate the safety and efficacy of SC PF-06801591 in patients with NSCLC or urothelial carcinoma as well as confirm the recommended Phase 2 dose.

DETAILED DESCRIPTION:
Protocol B8011001 is a Phase 1, two part, open-label, multi center, multiple-dose, safety, efficacy, PK, and PD study of PF-06801591 administered intravenously (IV) or subcutaneous (SC) in previously treated adult patients with locally advanced or metastatic melanoma, squamous cell carcinoma head and neck (SCCHN), ovarian carcinoma, sarcoma, non-small cell lung carcinoma (NSCLC), urothelial carcinoma or other solid tumors.

The first part of the study, Part 1 dose escalation, was designed to assess the safety and tolerability of increasing dose levels of IV or SC administered PF-06801591 to establish the maximum tolerated dose (MTD) using a modified Toxicity Probability Interval (mTPI) design. Part 2 expansion is designed to further evaluate the safety and efficacy of 300 mg of PF-06801591 administered SC once every 4 weeks in patients with NSCLC or urothelial carcinoma as well as confirm the recommended Phase 2 dose (RP2D). Part 1 enrollment has completed, enrollment will only be allowed for Part 2.

ELIGIBILITY:
Inclusion Criteria (Part 2 Only):

* Histological or cytological diagnosis of locally advanced or metastatic NSCLC or urothelial carcinoma who have progressed on or were intolerant to standard of care systemic therapy, or for whom standard of care systemic therapy was refused (refusal must be documented) or unavailable.
* No prior treatment with anti-PD-1 or anti-PD-L1 therapy.
* NSCLC patients whose tumor is not known to have ALK or EGFR mutations must have progressed on or after no more than 1 prior line of platinum-containing systemic therapy or were intolerant or refused standard of care systemic therapy.
* NSCLC patients whose tumor is known to have ALK or EGFR mutation must have received prior systemic therapies that only include 1 or more lines of ALK or EGFR targeting drugs and chemotherapy limited to 1 line of a platinum-based regimen and they must have progressed on or after both types of therapies.
* Urothelial carcinoma patients must have received up to 2 lines of prior systemic therapy and progressed on or after, experienced disease recurrence within 12 months of neoadjuvant or adjuvant treatment, were intolerant to, ineligible or refused platinum-containing systemic therapy. If urothelial cancer patients are treatment naïve and eligible for platinum-containing systemic therapy but are refusing platinum chemotherapy, they must also be documented to have previous PD-L1 high status.
* Provide archived tumor tissue sample taken within the past 2 years or provide a fresh tumor biopsy sample.
* At least one measurable lesion as defined by RECIST version 1.1.
* Adequate renal, liver, thyroid and bone marrow function.
* Performance status 0 or 1.
* Patient is capable of receiving study treatment for at least 8 weeks.

Exclusion Criteria (Part 2 Only)

* Active brain or leptomeningeal metastases.
* Active, known or suspected autoimmune disease. Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Diagnosis of prior immunodeficiency or organ transplant requiring immunosuppressive therapy or prior allogeneic bone marrow or hematopoietic stem cell transplant.
* Patients with a condition requiring systemic treatment with either corticosteroids (>10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patients with a history of interstitial lung disease, non-infectious pneumonitis, or active pulmonary tuberculosis. Those with active lung infections requiring treatment are also excluded.
* History of Grade ≥3 immune mediated AE (including AST/ALT elevations that where considered drug related and cytokine release syndrome) that was considered related to prior immune modulatory therapy (eg, immune checkpoint inhibitors, co-stimulatory agents, etc.) and required immunosuppressive therapy.
* Active hepatitis B or C, HIV/AIDS.
* Other potentially metastatic malignancy within past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (63):
- United States (21):
  - Clinical Research Unit, Los Angeles, California
  - Ronald Reagan Medical Center, Department of Radiological Sciences, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - UCLA Hematology & Oncology Clinic, Los Angeles, California
  - Santa Monica UCLA Hematology & Oncology Clinic, Santa Monica, California
  - Norton Cancer Institute, Multidisciplinary Clinic, Louisville, Kentucky
  - Norton Cancer Institute, Norton Healthcare Pavilion, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - University of Rochester, Rochester, New York
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
- Bulgaria (4):
  - MHAT Uni Hospital OOD, Panagyurishte, Pazardzhik
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - "MHAT for Women Health - Nadezhda" OOD, Sofia
  - SHATOD "Dr. Marko Antonov Markov - Varna" EOOD, Varna
- Malaysia (4):
  - Hospital Sultan Ismail, Johor Bahru, Johor
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Clinical Research Centre(Crc), Hospital Umum Sarawak, Kuching, Sarawak
- Poland (6):
  - Szpitale Pomorskie Sp. z.o.o., Oddzial Onkologii i Radioterapii, Gdynia
  - Regionalny Szpital Specjalistyczny im. dr. Wl. Bieganskiego w Grudziadzu, Grudziądz
  - Centrum Badan Klinicznych JCI Life Science Park, Krakow
  - Mazowiecki Szpital Specjalistyczny im. Dr. Jozefa Psarskiego w Ostrolece, Osrodek Onkologiczny, Ostrołęka
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Otwock
  - Centrum Onkologii-Instytut im.Marii Sklodowskiej-Curie, Warsaw
- Russia (10):
  - Sbhi "Lrcod", Vsevolozhsky District, Leningradskaya Oblast'
  - SBHI ¨Saint-Petersburg clinical scientific practical center of specialized types of, Pesochny Village, Sankt-Peterburg
  - SBHI "ChRCCO and NM", Chelyabinsk
  - MROI n.a. P.A. Gertsen, filiation of FSBI "NMRC of radiology" MoH Russia, Moscow
  - BHI of Omsk Region "Clinical Oncology Dispensary", Omsk
  - Joint Stock Company Current medical technologies, Saint Petersburg
  - Joint-Stock Company Current medical technologies, Saint Petersburg
  - Non-governmental Healthcare Institution ¨Railway Clinical Hospital of JSC ¨Russian Railways¨, Saint Petersburg
  - SPb SBHI "City Clinical Oncology Dispensary", Saint Petersburg
  - SBHI YaR ¨Regional clinical oncology hospital¨, Yaroslavl
- South Korea (9):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Division of Medical Oncology, Severance Hospital, Yonsei University Health System, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
- Ukraine (9):
  - Communal Non-profit Institution "City Clinical Hospital #4" of Dnipro City Council, Department of, Dnipro
  - Communal non-Commercial Enterprise "Prykarpatski Clinical Oncological Center of Ivano-, Ivano-Frankivsk
  - Grigoriev Radiological Institute of the National Academy of Medical Sciences of Ukraine,, Kharkiv
  - Communal Non-profit Institution of Kharkiv Regional Council "Regional Clinical Specialized Health, Kharkiv
  - "Specialized Clinic "Prognosis Optima" LLC, Kyiv
  - Communal noncommercial enterprise Sumy regional Rada Sumy regional clinical oncologic dispensary,, Sumy
  - Communal Non-profit Institution "Central City Clinical Hospital" of Uzhhorod City Council,, Uzhhorod
  - Vinnytsia Regional Clinical Oncological Hospital, Vinnytsia
  - Communal Institution ¨Zaporizhzhya Regional Clinical Oncological Dispensary¨, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Sako C, Duan C, Maresca K, Kent S, Schmidt TG, Aerts HJWL, Parikh RB, Simon GR, Jordan P. Real-World and Clinical Trial Validation of a Deep Learning Radiomic Biomarker for PD-(L)1 Immune Checkpoint Inhibitor Response in Advanced Non-Small Cell Lung Cancer. JCO Clin Cancer Inform. 2024 Dec;8:e2400133. doi: 10.1200/CCI.24.00133. Epub 2024 Dec 13. PMID 39671539
- [Derived] Hu-Lieskovan S, Braiteh F, Grilley-Olson JE, Wang X, Forgie A, Bonato V, Jacobs IA, Chou J, Johnson ML. Association of Tumor Mutational Burden and Immune Gene Expression with Response to PD-1 Blockade by Sasanlimab Across Tumor Types and Routes of Administration. Target Oncol. 2021 Nov;16(6):773-787. doi: 10.1007/s11523-021-00833-2. Epub 2021 Oct 25. PMID 34694529
- [Derived] Johnson ML, Braiteh F, Grilley-Olson JE, Chou J, Davda J, Forgie A, Li R, Jacobs I, Kazazi F, Hu-Lieskovan S. Assessment of Subcutaneous vs Intravenous Administration of Anti-PD-1 Antibody PF-06801591 in Patients With Advanced Solid Tumors: A Phase 1 Dose-Escalation Trial. JAMA Oncol. 2019 Jul 1;5(7):999-1007. doi: 10.1001/jamaoncol.2019.0836. PMID 31145415
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B8011001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 147 participants were enrolled in this study, and 146 participants received study treatment. For Part 1, 40 participants were enrolled and treated. For Part 2, 107 participants were enrolled including 68 participants with non small cell lung cancer (NSCLC) and 39 participants with urothelial carcinoma (UC), and 106 participants received study treatment.
Groups:
- Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]): Participants received PF-06801591 0.5 mg/kg IV every 3 weeks for 21-day cycles. (maximum of 1186 days)
- Part 1: PF-06801591 1 mg/kg (IV): Participants received PF-06801591 1 mg/kg IV every 3 weeks for 21-day cycles. (maximum of 659 days)
- Part 1: PF-06801591 3 mg/kg (IV): Participants received PF-06801591 3 mg/kg IV every 3 weeks for 21-day cycles. (maximum of 1606 days)
- Part 1: PF-06801591 10 mg/kg (IV): Participants received PF-06801591 10 mg/kg IV every 3 weeks for 21-day cycles. (maximum of 445 days)
- Part 1: PF-06801591 300 mg (Subcutaneously [SC]): Participants received PF-06801591 300 mg SC every 4 weeks for 28-day cycles. (maximum of 419 days)
- Part 2: PF-06801591 300 mg (SC) for NSCLC: Participants with NSCLC received PF-06801591 300 mg SC every 4 weeks for 28-day cycles. (maximum of 851 days)
- Part 2: PF-06801591 300 mg (SC) for UC: Participants with UC received PF- 06801591 300 mg SC every 4 weeks for 28-day cycles. (maximum of 841 days)
Period: Overall Study
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Started | 2 | 8 | 8 | 7 | 15 | 68 | 39
Treated | 2 | 8 | 8 | 7 | 15 | 68 | 38
Completed | 1 | 0 | 2 | 1 | 2 | 10 | 5
Not Completed | 1 | 8 | 6 | 6 | 13 | 58 | 34
Not completed — Death | 1 | 6 | 5 | 6 | 9 | 32 | 21
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Participant refused further follow-up | 0 | 2 | 1 | 0 | 3 | 20 | 7
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 4 | 5

BASELINE CHARACTERISTICS:
Population: Baseline population included all enrolled participants who received at least 1 dose of study treatment. One participant who enrolled in Part 2: PF-06801591 300 mg (SC) for UC arm was not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC | Total
Number analyzed (Participants) | 2 | 8 | 8 | 7 | 15 | 68 | 38 | 146
Age, Customized [Number; unit: Participants]
  18-44 Years | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 4
  45-64 Years | 1 | 3 | 5 | 3 | 10 | 28 | 16 | 66
  >=65 Years | 1 | 5 | 2 | 3 | 5 | 39 | 21 | 76
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 5 | 4 | 11 | 15 | 13 | 56
  Male | 0 | 2 | 3 | 3 | 4 | 53 | 25 | 90
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 2 | 7 | 7 | 4 | 12 | 50 | 30 | 112
  Black or African American | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3
  Asian | 0 | 0 | 0 | 2 | 1 | 18 | 8 | 29
  Other | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose-Limiting Toxicities (DLT) - Part 1
Description: DLT was defined as any of the following drug-related adverse events (AEs) occurring during the first cycle (21 days for IV dosing, 28 days for SC dosing) in Part 1: Grade 5 AE; Grade 4 neutropenia lasting >5 days from initiation of granulocyte colony stimulating factor; Grade 4 thrombocytopenia with bleeding; Platelet transfusion requirement or a platelet count <10,000/uL; Grade 4 non-hematologic AE; Grade 3 AE lasting >7 days despite optimal supportive care; Grade 3 central nervous system AE regardless of duration; met criteria for drug induced liver injury. Severity of AEs were graded according to Common Terminology Criteria for Adverse Events (CTCAE) v4.03. Grade 3 = severe AE. Grade 4 = life-threatening consequences; urgent intervention indicated. Grade 5 = death related to AE.
Time Frame: Cycle 1 in Part 1 (21 days for IV administration of PF-06801591; 28 days for SC administration of PF-06801591)
Population: DLT analysis population included all enrolled participants who received at least 1 dose of study treatment and who did not have major treatment deviations during Cycle 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC])
Number analyzed (Participants) | 2 | 8 | 8 | 7 | 15
Percentage of Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With All-Causality Treatment-Emergent Adverse Events (AEs) - Part 1 and Part 2
Description: AE = any untoward medical occurrence in participant who received study treatment without regard to possibility of causal relationship. Treatment-emergent events = between first dose of study treatment and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Grades of severity were defined by CTCAE v4.03. Grades of severity were defined by CTCAE v4.03. Grade 3 = severe AE. Grade 4 = life-threatening consequences; urgent intervention indicated. Grade 5 = death related to AE.
Time Frame: Baseline up to 28 days after last dose of study treatment (maximum of 1634 days)
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 2 | 8 | 8 | 7 | 15 | 68 | 38
Participants
  Participants with AEs | 2 | 7 | 8 | 7 | 15 | 62 | 36
  Participants with SAEs | 1 | 3 | 3 | 3 | 3 | 18 | 13
  Participants with maximum Grade 3 or 4 AEs | 2 | 2 | 3 | 2 | 4 | 18 | 13
  Participants with maximum Grade 5 AEs | 0 | 1 | 1 | 2 | 0 | 8 | 5

3. Primary Outcome: Number of Participants With Treatment-Related Treatment-Emergent Adverse Events (AEs) - Part 1 and Part 2
Description: Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Treatment-emergent events = between first dose of study treatment and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-related AEs and SAEs were determined by the investigator. Grades of severity were defined by CTCAE v4.03. Grades of severity were defined by CTCAE v4.03. Grade 3 = severe AE. Grade 4 = life-threatening consequences; urgent intervention indicated. Grade 5 = death related to AE.
Time Frame: Baseline up to 28 days after last dose of study treatment (maximum of 1634 days)
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 2 | 8 | 8 | 7 | 15 | 68 | 38
Participants
  Participants with AEs | 2 | 6 | 7 | 6 | 13 | 42 | 17
  Participants with SAEs | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Participants with maximum of Grade 3 or 4 AEs | 1 | 1 | 1 | 1 | 1 | 9 | 5
  Participants with maximum of Grade 5 AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Laboratory Test Abnormalities - Part 1 and Part 2
Description: Following parameters were analyzed for laboratory examination: hematology (anemia, hemoglobin increased, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, white blood cell decreased); chemistries (increase of alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, blood bilirubin, CPK, creatinine, gamma-glutamyl transferase [GGT], lipase, and serum amylase); urinalysis (proteinuria); coagulation (activated partial thromboplastin time prolonged, international normalized ratio [INR] increased). Grades of severity were defined by CTCAE v4.03. Grade 0 = No Change from normal or reference range (this grade is not included in the CTCAE v4.03 document but may used in certain circumstances). Grade 1 = mild adverse event (AE). Grade 2 = moderate AE; Grade 3 = severe AE. Grade 4 = life-threatening consequences; urgent intervention indicated. Grade 5 = death related to AE.
Time Frame: Baseline up to 28 days after last dose of study treatment (maximum of 1634 days)
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 2 | 7 | 8 | 7 | 15 | 68 | 38
Participants
  ANEMIA: Grade 0 | 0 | 2 | 1 | 1 | 1 | 16 | 6
  ANEMIA: Grade 1 | 1 | 1 | 4 | 5 | 5 | 38 | 16
  ANEMIA: Grade 2 | 1 | 4 | 3 | 1 | 8 | 13 | 9
  ANEMIA: Grade 3 | 0 | 0 | 0 | 0 | 1 | 1 | 7
  ANEMIA: Grade 4 | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  HEMOGLOBIN INCREASED: Grade 0 | 2 | 7 | 8 | 7 | 15 | 60 | 35
  HEMOGLOBIN INCREASED: Grade 1 | 0 | 0 | 0 | 0 | 0 | 7 | 3
  HEMOGLOBIN INCREASED: Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  HEMOGLOBIN INCREASED: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HEMOGLOBIN INCREASED: Grade 4 | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  LYMPHOCYTE COUNT DECREASED: Grade 0 | 0 | 3 | 0 | 1 | 9 | 27 | 20
  LYMPHOCYTE COUNT DECREASED: Grade 1 | 0 | 0 | 2 | 1 | 2 | 21 | 11
  LYMPHOCYTE COUNT DECREASED: Grade 2 | 2 | 2 | 6 | 4 | 1 | 15 | 5
  LYMPHOCYTE COUNT DECREASED: Grade 3 | 0 | 1 | 0 | 1 | 3 | 5 | 2
  LYMPHOCYTE COUNT DECREASED: Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  LYMPHOCYTE COUNT INCREASED: Grade 0 | 2 | 7 | 8 | 7 | 14 | 63 | 37
  LYMPHOCYTE COUNT INCREASED: Grade 1 | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  LYMPHOCYTE COUNT INCREASED: Grade 2 | 0 | 0 | 0 | 0 | 1 | 5 | 1
  LYMPHOCYTE COUNT INCREASED: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMPHOCYTE COUNT INCREASED: Grade 4 | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  NEUTROPHIL COUNT DECREASED: Grade 0 | 2 | 6 | 7 | 5 | 13 | 61 | 35
  NEUTROPHIL COUNT DECREASED: Grade 1 | 0 | 1 | 1 | 2 | 1 | 4 | 0
  NEUTROPHIL COUNT DECREASED: Grade 2 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  NEUTROPHIL COUNT DECREASED: Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  NEUTROPHIL COUNT DECREASED: Grade 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  PLATELET COUNT DECREASED: Grade 0 | 1 | 7 | 7 | 6 | 12 | 56 | 33
  PLATELET COUNT DECREASED: Grade 1 | 1 | 0 | 1 | 1 | 3 | 12 | 5
  PLATELET COUNT DECREASED: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLATELET COUNT DECREASED: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLATELET COUNT DECREASED: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WHITE BLOOD CELL DECREASED: Grade 0 | 1 | 5 | 5 | 3 | 10 | 62 | 34
  WHITE BLOOD CELL DECREASED: Grade 1 | 1 | 1 | 3 | 4 | 4 | 5 | 3
  WHITE BLOOD CELL DECREASED: Grade 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  WHITE BLOOD CELL DECREASED: Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  WHITE BLOOD CELL DECREASED: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALANINE AMINOTRANSFERASE INCREASED: Grade 0 | 2 | 7 | 8 | 4 | 14 | 45 | 31
  ALANINE AMINOTRANSFERASE INCREASED: Grade 1 | 0 | 0 | 0 | 3 | 1 | 19 | 3
  ALANINE AMINOTRANSFERASE INCREASED: Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  ALANINE AMINOTRANSFERASE INCREASED: Grade 3 | 0 | 0 | 0 | 0 | 0 | 3 | 1
  ALANINE AMINOTRANSFERASE INCREASED: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALKALINE PHOSPHATASE INCREASED: Grade 0 | 1 | 4 | 5 | 4 | 6 | 36 | 21
  ALKALINE PHOSPHATASE INCREASED: Grade 1 | 0 | 2 | 3 | 2 | 7 | 22 | 11
  ALKALINE PHOSPHATASE INCREASED: Grade 2 | 1 | 1 | 0 | 0 | 2 | 7 | 4
  ALKALINE PHOSPHATASE INCREASED: Grade 3 | 0 | 0 | 0 | 1 | 0 | 3 | 2
  ALKALINE PHOSPHATASE INCREASED: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ASPARTATE AMINOTRANSFERASE INCREASED: number analyzed (Participants) | 2 | 7 | 8 | 7 | 15 | 67 | 38
  ASPARTATE AMINOTRANSFERASE INCREASED: Grade 0 | 0 | 5 | 7 | 5 | 11 | 44 | 23
  ASPARTATE AMINOTRANSFERASE INCREASED: Grade 1 | 2 | 2 | 1 | 1 | 4 | 17 | 13
  ASPARTATE AMINOTRANSFERASE INCREASED: Grade 2 | 0 | 0 | 0 | 0 | 0 | 5 | 1
  ASPARTATE AMINOTRANSFERASE INCREASED: Grade 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  ASPARTATE AMINOTRANSFERASE INCREASED: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  BLOOD BILIRUBIN INCREASED: Grade 0 | 1 | 7 | 7 | 6 | 13 | 58 | 34
  BLOOD BILIRUBIN INCREASED: Grade 1 | 0 | 0 | 1 | 0 | 1 | 6 | 3
  BLOOD BILIRUBIN INCREASED: Grade 2 | 1 | 0 | 0 | 0 | 1 | 3 | 1
  BLOOD BILIRUBIN INCREASED: Grade 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  BLOOD BILIRUBIN INCREASED: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CPK INCREASED: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 0
  CPK INCREASED: Grade 0 |  |  |  |  |  | 3 |
  CPK INCREASED: Grade 1 |  |  |  |  |  | 0 |
  CPK INCREASED: Grade 2 |  |  |  |  |  | 0 |
  CPK INCREASED: Grade 3 |  |  |  |  |  | 0 |
  CPK INCREASED: Grade 4 |  |  |  |  |  | 0 |
  CREATININE INCREASED: Grade 0 | 0 | 0 | 3 | 0 | 13 | 58 | 2
  CREATININE INCREASED: Grade 1 | 1 | 6 | 4 | 7 | 1 | 6 | 30
  CREATININE INCREASED: Grade 2 | 1 | 1 | 1 | 0 | 1 | 3 | 5
  CREATININE INCREASED: Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  CREATININE INCREASED: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GGT INCREASED: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 4 | 2
  GGT INCREASED: Grade 0 | 0 |  |  |  |  | 0 | 0
  GGT INCREASED: Grade 1 | 1 |  |  |  |  | 2 | 1
  GGT INCREASED: Grade 2 | 0 |  |  |  |  | 1 | 0
  GGT INCREASED: Grade 3 | 0 |  |  |  |  | 1 | 1
  GGT INCREASED: Grade 4 | 0 |  |  |  |  | 0 | 0
  HYPERCALCEMIA: Grade 0 | 2 | 7 | 8 | 7 | 13 | 51 | 31
  HYPERCALCEMIA: Grade 1 | 0 | 0 | 0 | 0 | 1 | 15 | 5
  HYPERCALCEMIA: Grade 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  HYPERCALCEMIA: Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  HYPERCALCEMIA: Grade 4 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  HYPERGLYCEMIA: Grade 0 | 2 | 5 | 8 | 6 | 14 | 24 | 12
  HYPERGLYCEMIA: Grade 1 | 0 | 0 | 0 | 0 | 0 | 31 | 21
  HYPERGLYCEMIA: Grade 2 | 0 | 0 | 0 | 0 | 0 | 10 | 4
  HYPERGLYCEMIA: Grade 3 | 0 | 2 | 0 | 0 | 1 | 3 | 1
  HYPERGLYCEMIA: Grade 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  HYPERKALEMIA: Grade 0 | 2 | 6 | 7 | 7 | 15 | 48 | 27
  HYPERKALEMIA: Grade 1 | 0 | 0 | 1 | 0 | 0 | 8 | 6
  HYPERKALEMIA: Grade 2 | 0 | 0 | 0 | 0 | 0 | 11 | 3
  HYPERKALEMIA: Grade 3 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  HYPERKALEMIA: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPERMAGNESEMIA: Grade 0 | 1 | 7 | 7 | 5 | 15 | 55 | 35
  HYPERMAGNESEMIA: Grade 1 | 1 | 0 | 1 | 2 | 0 | 6 | 3
  HYPERMAGNESEMIA: Grade 2 | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  HYPERMAGNESEMIA: Grade 3 | 0 | 0 | 0 | 0 | 0 | 7 | 0
  HYPERMAGNESEMIA: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPERNATREMIA: Grade 0 | 2 | 5 | 8 | 6 | 13 | 51 | 35
  HYPERNATREMIA: Grade 1 | 0 | 2 | 0 | 1 | 2 | 8 | 2
  HYPERNATREMIA: Grade 2 | 0 | 0 | 0 | 0 | 0 | 7 | 0
  HYPERNATREMIA: Grade 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  HYPERNATREMIA: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  HYPOALBUMINEMIA: Grade 0 | 1 | 5 | 5 | 3 | 10 | 40 | 23
  HYPOALBUMINEMIA: Grade 1 | 0 | 2 | 2 | 4 | 2 | 18 | 11
  HYPOALBUMINEMIA: Grade 2 | 1 | 0 | 1 | 0 | 2 | 10 | 4
  HYPOALBUMINEMIA: Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  HYPOALBUMINEMIA: Grade 4 | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  HYPOCALCEMIA: Grade 0 | 1 | 6 | 5 | 5 | 13 | 49 | 30
  HYPOCALCEMIA: Grade 1 | 1 | 1 | 3 | 2 | 1 | 12 | 7
  HYPOCALCEMIA: Grade 2 | 0 | 0 | 0 | 0 | 1 | 7 | 0
  HYPOCALCEMIA: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPOCALCEMIA: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  HYPOGLYCEMIA: Grade 0 | 2 | 7 | 8 | 7 | 15 | 60 | 32
  HYPOGLYCEMIA: Grade 1 | 0 | 0 | 0 | 0 | 0 | 8 | 6
  HYPOGLYCEMIA: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPOGLYCEMIA: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPOGLYCEMIA: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPOKALEMIA: Grade 0 | 1 | 7 | 5 | 6 | 10 | 61 | 33
  HYPOKALEMIA: Grade 1 | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  HYPOKALEMIA: Grade 2 | 1 | 0 | 3 | 1 | 4 | 7 | 3
  HYPOKALEMIA: Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  HYPOKALEMIA: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPOMAGNESEMIA: Grade 0 | 2 | 6 | 7 | 7 | 8 | 42 | 29
  HYPOMAGNESEMIA: Grade 1 | 0 | 1 | 1 | 0 | 5 | 14 | 8
  HYPOMAGNESEMIA: Grade 2 | 0 | 0 | 0 | 0 | 2 | 8 | 1
  HYPOMAGNESEMIA: Grade 3 | 0 | 0 | 0 | 0 | 0 | 4 | 0
  HYPOMAGNESEMIA: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPONATREMIA: Grade 0 | 0 | 4 | 7 | 5 | 8 | 45 | 25
  HYPONATREMIA: Grade 1 | 0 | 2 | 1 | 1 | 5 | 19 | 10
  HYPONATREMIA: Grade 2 | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  HYPONATREMIA: Grade 3 | 2 | 0 | 0 | 1 | 2 | 3 | 2
  HYPONATREMIA: Grade 4 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  HYPOPHOSPHATEMIA: number analyzed (Participants) | 2 | 7 | 8 | 7 | 15 | 67 | 38
  HYPOPHOSPHATEMIA: Grade 0 | 1 | 5 | 6 | 7 | 15 | 56 | 27
  HYPOPHOSPHATEMIA: Grade 1 | 0 | 0 | 0 | 0 | 0 | 3 | 7
  HYPOPHOSPHATEMIA: Grade 2 | 1 | 2 | 2 | 0 | 0 | 7 | 4
  HYPOPHOSPHATEMIA: Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  HYPOPHOSPHATEMIA: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LIPASE INCREASED: number analyzed (Participants) | 2 | 7 | 8 | 7 | 15 | 68 | 37
  LIPASE INCREASED: Grade 0 | 2 | 4 | 5 | 7 | 13 | 50 | 23
  LIPASE INCREASED: Grade 1 | 0 | 3 | 1 | 0 | 0 | 11 | 7
  LIPASE INCREASED: Grade 2 | 0 | 0 | 1 | 0 | 0 | 4 | 3
  LIPASE INCREASED: Grade 3 | 0 | 0 | 1 | 0 | 1 | 1 | 3
  LIPASE INCREASED: Grade 4 | 0 | 0 | 0 | 0 | 1 | 2 | 1
  SERUM AMYLASE INCREASED: Grade 0 | 1 | 6 | 7 | 6 | 13 | 45 | 23
  SERUM AMYLASE INCREASED: Grade 1 | 1 | 1 | 1 | 0 | 1 | 16 | 10
  SERUM AMYLASE INCREASED: Grade 2 | 0 | 0 | 0 | 1 | 0 | 4 | 2
  SERUM AMYLASE INCREASED: Grade 3 | 0 | 0 | 0 | 0 | 1 | 3 | 3
  SERUM AMYLASE INCREASED: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PROTEINURIA: number analyzed (Participants) | 2 | 7 | 8 | 6 | 15 | 66 | 38
  PROTEINURIA: Grade 0 | 0 | 5 | 4 | 1 | 9 | 46 | 15
  PROTEINURIA: Grade 1 | 1 | 2 | 3 | 3 | 6 | 15 | 17
  PROTEINURIA: Grade 2 | 1 | 0 | 1 | 2 | 0 | 5 | 5
  PROTEINURIA: Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  PROTEINURIA: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED: Grade 0 | 1 | 6 | 5 | 4 | 11 | 44 | 19
  ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED: Grade 1 | 1 | 1 | 3 | 3 | 4 | 19 | 15
  ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED: Grade 2 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED: Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED: Grade 4 | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.
  INR INCREASED: number analyzed (Participants) | 2 | 7 | 8 | 7 | 15 | 68 | 36
  INR INCREASED: Grade 0 | 2 | 5 | 6 | 4 | 12 | 39 | 31
  INR INCREASED: Grade 1 | 0 | 2 | 1 | 3 | 3 | 25 | 4
  INR INCREASED: Grade 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  INR INCREASED: Grade 3 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  INR INCREASED: Grade 4 | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined. | NA — CTCAE grade not defined.

5. Primary Outcome: Objective Response Rate (ORR) Based on RECIST Version 1.1 - Part 2
Description: ORR was defined as percentage of participants with confirmed objective response (OR) of complete response (CR) and partial response (PR) based on RECIST version 1.1. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis < 10 mm). All target lesions must be assessed. PR was defined as >= 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. All target lesions must be assessed.
Time Frame: Baseline up to end of treatment in Part 2 (maximum of 851 days)
Population: Analysis population included all the randomized participants who received at least 1 dose of study medication, had measurable disease baseline assessment (within 28 days prior to study entry) and at least 1 post baseline assessment or disease progression, global deterioration of health status, or death.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 67 | 38
Percentage | 16.4 [8.5 to 27.5] | 18.4 [7.7 to 34.3]

6. Primary Outcome: Objective Response Rate (ORR) Based on Immune Related RECIST (irRECIST) - Part 2
Description: ORR was defined as percentage of participants with objective response (OR) of complete response (CR) and partial response (PR) based on irRECIST. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis < 10 mm). All target lesions must be assessed. PR was defined as >= 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. All target lesions must be assessed.
Time Frame: Baseline up to end of treatment in Part 2 (maximum of 851 days)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 67 | 38
Percentage of Participants | 19.4 [10.8 to 30.9] | 21.1 [9.6 to 37.3]

7. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-06801591 - Part 1
Description: Cmax was the maximum concentration after dose administration observed directly from the data.
Time Frame: Pre-dose, 1 and 24 hours post dose on Cycle 1 Day 1, and pre-dose and 1 hour post dose on Cycle 4 Day 1 in Part 1
Population: Analysis population included all enrolled participants treated who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC])
Number analyzed (Participants) | 2 | 8 | 8 | 7 | 15
ug/mL
  Cycle 1 Day 1 | NA (NA) — Geometric mean and geometric coefficient of variation were not reported for n < 3. | 21.52 (23) | 69.63 (28) | 217.2 (36) | 21.24 (50)
  Cycle 4 Day 1 | NA (NA) — Geometric mean and geometric coefficient of variation were not reported for n < 3. | 30.10 (16) | 86.34 (52) | 402.6 (42) | 56.48 (29)

8. Secondary Outcome: AUClast of PF-06801591 in Part 1.
Description: Area Under the Concentration Versus Time Curve (AUC) From Time Zero to the Last Quantifiable Time Point Prior to the Next Dose (AUClast) of PF-06801591 - Part 1
Time Frame: Pre-dose, 1 and 24 hours post dose on Cycle 1 Day 1 in Part 1
Population: Analysis population included all enrolled participants treated who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC])
Number analyzed (Participants) | 2 | 7 | 7 | 7 | 15
ug*hr/mL | NA (NA) — Geometric mean and geometric coefficient of variation were not reported for n < 3. | 4700 (41) | 14770 (27) | 46780 (49) | 9923 (65)

9. Secondary Outcome: Clearance (CL) of PF-06801591 - Part 1
Description: CL for IV dosing. CL was calculated by dose / AUCtau for Cycles 1 and 4 IV dosing. AUCtau was defined as area under the serum concentration time profile from time zero to time tau, the dosing interval, where tau = 504 hours for every 3 weeks (Q3W) IV dosing reporting arm.
Time Frame: Pre-dose, 1 and 24 hours post dose on Cycle 1 Day 1, and pre-dose and 1 hour post dose on Cycle 4 Day 1 in Part 1
Population: Analysis population included all enrolled participants treated who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV)
Number analyzed (Participants) | 2 | 2 | 3 | 4
L/hr
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Cycle 1 Day 1 |  | NA (NA) — Geometric mean and geometric coefficient of variation were not reported for n < 3. |  |
  Cycle 4 Day 1 | NA (NA) — Geometric mean and geometric coefficient of variation were not reported for n < 3. | NA (NA) — Geometric mean and geometric coefficient of variation were not reported for n < 3. | 0.006045 (57) | 0.004984 (14)

10. Secondary Outcome: Volume of Distribution at Steady State (Vss) of PF-06801591 - Part 1
Description: Steady state volume of distribution of PF-0680159 for IV dosing. Vss was calculated by CL*MRT. CL was the clearance for IV dosing. MRT was the mean residence time calculated for a single IV dose as AUMCinf/AUCinf - (DOF/2). AUMCinf was the area under the moment curve from time 0 extrapolated to infinity. DOF was the duration of infusion. AUCinf was the area under the serum concentration time profile from time 0 extrapolated to infinity.
Time Frame: Pre-dose, 1 and 24 hours post dose on Cycle 1 Day 1, and pre-dose and 1 hour post dose on Cycle 4 Day 1 in Part 1
Population: The PK parameter analysis population was defined as all enrolled participants in Part 1 who received study drug following IV administration and had sufficient information to estimate at least 1 of the pharmacokinetic (PK) parameters of interest. Number of participants analyzed represents the total number of participants in each treatment group in the PK parameter analysis population. Number analyzed represents the number of participants who had reportable parameter values of Vss.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV)
Number analyzed (Participants) | 2 | 8 | 8 | 7
L
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Cycle 1 Day 1 |  | NA (NA) — Geometric mean and geometric coefficient of variation were not reported for n < 3. |  |
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Accumulation Ratio (Rac) of PF-06801591 - Part 1
Description: Rac was calculated by (Cycle 4 AUCtau) / (Cycle 1 AUCtau). AUCtau was Area under the serum concentration time profile from time zero to time tau, the dosing interval, where tau = 504 hours for Q3W IV dosing and tau = 672 hours for every 4 weeks (Q4W) SC dosing.
Time Frame: Pre-dose and 1 hour post dose on Day 1 of Cycles 1 and 4 in Part 1
Population: Analysis population included all enrolled participants treated who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC])
Number analyzed (Participants) | 2 | 2 | 2 | 4 | 3
Ratio | NA (NA) — Geometric mean and geometric coefficient of variation were not reported for n < 3. | NA (NA) — Geometric mean and geometric coefficient of variation were not reported for n < 3. | NA (NA) — Geometric mean and geometric coefficient of variation were not reported for n < 3. | 2.360 (12) | 2.073 (31)

12. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of PF-06801591 - Part 1
Description: t1/2 was calculated by Loge(2)/kel. kel was the terminal phase rate constant calculated by a linear regression of the log linear concentration time curve. Only those data points judged to describe the terminal log linear decline were used in the regression.
Time Frame: Pre-dose and 1 hour post dose on Day 1 of Cycles 1 and 4 in Part 1
Population: The PK parameter analysis population was defined as all enrolled participants in Part 1 who received study drug following IV or SC administration and had sufficient information to estimate at least 1 of the PK parameters of interest. Number of participants analyzed represents the total number of participants in each treatment group in the PK parameter analysis population. Number analyzed represents the number of participants who had reportable parameter values of t1/2.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC])
Number analyzed (Participants) | 2 | 8 | 8 | 7 | 15
Days
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Cycle 1 Day 1 |  | NA (NA) — Mean and standard deviation were not reported for n<3. |  |  |
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Cycle 4 Day 1 |  |  |  |  | NA (NA) — Mean and standard deviation were not reported for n<3.

13. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Against PF-06801591 - Part 1 and Part 2
Description: Number of participants with ADA positive against PF-06801591 after IV and SC dosing - Part 1 and Part 2. A participant was ADA positive if (1) baseline titer was missing or negative and participant had ≥ 1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a ≥ 0.602 in titer from baseline in ≥ 1 post-treatment sample (treatment-boosted). Participants who were ADA positive at baseline but did not become boosted post-treatment were considered as ADA negative.
Time Frame: Baseline up to end of treatment (maximum of 851 days)
Population: Analysis population included all participants who received at least 1 dose of study treatment and had at least 1 post-treatment ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV)
Number analyzed (Participants) | 14 | 64 | 37 | 2 | 6 | 7 | 6
Participants | 1 | 5 | 3 | 1 | 1 | 0 | 0

14. Secondary Outcome: Number of Participants With Neutralizing Antibodies (NAb) Positive Against PF-06801591 - Part 1 and Part 2
Description: Number of participants with NAb positive against PF-06801591 after IV and SC dosing - Part 1 and Part 2. A participant was NAb positive if (1) baseline titer was missing or negative and participant had ≥ 1 post-treatment positive titer (treatment-induced), or (2) positive titer at baseline and had a ≥ 0.602 in titer from baseline in ≥ 1 post-treatment sample (treatment-boosted). Participants who were NAb positive at baseline but did not become boosted post-treatment were considered as NAb negative.
Time Frame: Baseline up to end of treatment (maximum of 851 days)
Population: Analysis population included all participants who received at least 1 dose of study treatment and had at least 1 post-treatment ADA result. NAb-negative participants included participants who were ADA negative or ADA-positive participants who tested negative in the NAb assay.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV)
Number analyzed (Participants) | 14 | 64 | 37 | 2 | 6 | 7 | 6
Participants | 0 | 3 | 1 | 0 | 0 | 0 | 0

15. Secondary Outcome: Percentage of Baseline PD-1 Receptor Occupancy (RO) by PF-06801591 - Part 1
Description: PD-1 RO by sasanlimab was measured by the reduction of free receptor on the surface of CD8+ effector cells (CD3+, CD4-, CD8+, CD45RA+, CCR7-, CD279+) and CD8+ effector memory cells (CD3+, CD4-, CD8+, CD45RA-, CCR7-, CD279+) presented in pre- and postdose whole blood samples by flow cytometry. Percentage of baseline (ie, normalized change from baseline) PD-1 RO were calculated as [(percentage of cells at Cycle X Day X)/(percentage of cells at baseline)]*100, and are reported for this outcome measure. Baseline was defined as the most recent non-missing value prior to dosing.
Time Frame: Baseline, Days 1, 8, 15, 21 of Cycle 1, Day 1 of Cycles 2, 3, 5, Days 1, 15, 21 of Cycle 4, and end of treatment (EOT) in Part 1 (cycle = 21 days for IV dosing; cycle = 28 days for SC dosing)
Population: Analysis population included all enrolled participants with at least 1 of the pharmacodynamic/biomarker parameters evaluated at pre- and/or post dose.
Measure: Median (Full Range); unit: Percentage of Baseline
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC])
Number analyzed (Participants) | 2 | 8 | 7 | 7 | 15
Percentage of Baseline
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 8 | 7 | 6 | 13
  Cycle 1 Day 1 | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.1] | 0.56 [0.0 to 4.0] | 0.02 [0.0 to 0.6] | 0.32 [0.0 to 3.0]
  Cycle 1 Day 8: number analyzed (Participants) | 2 | 6 | 6 | 7 | 15
  Cycle 1 Day 8 | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.2] | 0.00 [0.0 to 1.4] | 0.00 [0.0 to 3.1]
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 6 | 7 | 7 | 12
  Cycle 1 Day 15 | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 1.3] | 0.00 [0.0 to 0.6] | 0.00 [0.0 to 7.7] | 0.57 [0.0 to 4.5]
  Cycle 1 Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13
  Cycle 1 Day 21 |  |  |  |  | 0.00 [0.0 to 1.0]
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 6 | 5 | 5 | 14
  Cycle 2 Day 1 | 1.48 [0.0 to 3.0] | 0.04 [0.0 to 1.7] | 0.82 [0.0 to 3.0] | 0.00 [0.0 to 1.0] | 0.00 [0.0 to 4.7]
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 4 | 6 | 5 | 11
  Cycle 3 Day 1 | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.2] | 0.47 [0.0 to 3.1] | 0.00 [0.0 to 2.3] | 0.00 [0.0 to 4.7]
  Cycle 4 Day 1: number analyzed (Participants) | 2 | 8 | 5 | 6 | 7
  Cycle 4 Day 1 | 0.80 [0.5 to 1.1] | 0.00 [0.0 to 0.0] | 0.05 [0.0 to 23.2] | 0.00 [0.0 to 2.1] | 0.00 [0.0 to 2.1]
  Cycle 4 Day 15: number analyzed (Participants) | 2 | 3 | 2 | 7 | 6
  Cycle 4 Day 15 | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 2.6] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.7] | 0.00 [0.0 to 1.4]
  Cycle 4 Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5
  Cycle 4 Day 21 |  |  |  |  | 1.31 [0.0 to 1.4]
  Cycle 5 Day 1: number analyzed (Participants) | 2 | 4 | 5 | 5 | 15
  Cycle 5 Day 1 | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 3.2] | 0.00 [0.0 to 1.2] | 0.00 [0.0 to 1.5]
  EOT: number analyzed (Participants) | 0 | 6 | 4 | 4 | 10
  EOT |  | 0.00 [0.0 to 0.5] | 0.00 [0.0 to 0.7] | 0.00 [0.0 to 0.5] | 0.17 [0.0 to 2.7]

16. Secondary Outcome: Number of Participants Achieving Objective Response (OR) Based on RECIST Version 1.1 - Part 1
Description: Number of participants achieving confirmed OR based on RECIST version 1.1 in Part 1. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis < 10 mm). All target lesions must be assessed. PR was defined as >= 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. All target lesions must be assessed.
Time Frame: Baseline up to end of treatment in Part 1 (maximum of 1606 days)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC])
Number analyzed (Participants) | 2 | 7 | 8 | 7 | 15
Participants | 1 | 2 | 1 | 2 | 1

17. Secondary Outcome: Number of Participants Achieving Objective Response (OR) Based on irRECIST - Part 1
Description: Number of participants achieving confirmed OR based on irRECIST in Part 1. OR = irCR + irPR. Overall immune related complete response (irCR) was defined as complete disappearance of all lesions (whether measurable or not) and no new lesions. All measurable lymph nodes also must have a reduction in short axis to <10 mm. Overall immune related partial response (irPR) was defined as sum of the diameters (longest for non nodal lesions, shortest for nodal lesions) of target and new measurable lesions decreases >=30%.
Time Frame: Baseline up to end of treatment in Part 1 (maximum of 1606 days)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC])
Number analyzed (Participants) | 2 | 7 | 8 | 7 | 15
Participants | 1 | 2 | 1 | 2 | 1

18. Secondary Outcome: Progression-Free Survival (PFS) Based on RECIST Version 1.1 and irRECIST - Part 1 and Part 2
Description: PFS was defined as the time from initiation of study intervention to first documentation of tumor progression or to death due to any cause, whichever occurred first. PFS was analyzed by the Kaplan-Meier approach for each tumor type. As this outcome measure was a secondary endpoint defined in the protocol to investigate preliminary signal of efficacy, the results were analyzed and are reported for Part 1 dose-escalation groups combined to provide more statistically meaningful results, instead of results analyzed by dose level with very limited number of participants in each group.
Time Frame: Baseline up to end of treatment (maximum of 1606 days)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Part 1: PF-06801591 0.5-10 mg/kg (Intravenously [IV]): This was a combined group of PF-06801591 0.5, 1, 3, and 10 mg/kg (IV) in Part 1. Participants received PF-06801591 0.5, 1, 3, or 10 mg/kg IV every 3 weeks for 21-day cycles. (up to a maximum of 233 weeks).
Arm/Group | Part 1: PF-06801591 0.5-10 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 24 | 15 | 67 | 38
Months
  RECIST v1.1 | 4.7 [1.4 to 8.3] | 3.0 [1.6 to 6.0] | 3.7 [1.9 to 5.5] | 2.9 [1.9 to 3.8]
  irRECIST | 4.9 [1.4 to 13.8] | 4.5 [1.9 to 13.7] | 5.5 [2.8 to 8.2] | 3.8 [2.0 to 14.5]

19. Secondary Outcome: Duration of Stable Disease (DOSD) Based on RECIST Version 1.1 and irRECIST - Part 1 and Part 2
Description: DOSD was analyzed by the Kaplan-Meier approach for each tumor type. Stable disease (SD) was defined as not qualifying for complete response (CR), partial response (PR), or progression. All target lesions must have been assessed. Stable could follow PR only in the rare case that the sum increased by less than 20% from the nadir, but enough that a previously documented 30% decrease no longer held. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must have decreased to normal size (short axis < 10 mm). All target lesions must have been assessed. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. All target lesions must have been assessed.
Time Frame: Baseline up to end of treatment (maximum of 1606 days)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 5 | 24 | 12
Months
  RECIST v1.1 | NA — Not estimable for n<2. | NA [4.6 to NA] — Not estimable for n<2. | 24.3 [13.8 to 34.9] | 5.7 [2.5 to 8.8] | 6.0 [3.8 to 7.3] | 6.5 [3.7 to 10.1] | 8.5 [3.7 to NA] — Not estimable.
  irRECIST | NA — Not estimable for n<2. | NA [4.6 to NA] — Not estimable for n<2. | 29.0 [20.0 to 37.9] | 5.7 [2.5 to 8.8] | 13.7 [3.3 to 13.7] | 7.5 [5.4 to 18.4] | 14.5 [3.7 to NA] — Not estimable.

20. Secondary Outcome: Duration of Response (DOR) Based on RECIST Version 1.1 and irRECIST - Part 1 and Part 2
Description: DOR was defined as the time from start date (which was the date of first documentation of PR or CR) to date of first documentation of objective progression or death. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. Objective progression was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm. As this outcome measure was a secondary endpoint defined in the protocol to investigate preliminary signal of efficacy, the results were analyzed and are reported for Part 1 dose-escalation groups combined to provide more statistically meaningful results, instead of results analyzed by dose level with very limited number of participants in each group.
Time Frame: Baseline up to end of treatment (maximum of 1606 days)
Population: Analysis population included all the randomized participants who received at least 1 dose of study medication, had measurable disease baseline assessment (within 28 days prior to study entry) and at least 1 post baseline assessment or disease progression, global deterioration of health status, or death. DOR was only applicable to those participants with an objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1: PF-06801591 0.5-10 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 6 | 1 | 13 | 8
Months
  RECIST v1.1: number analyzed (Participants) | 6 | 1 | 11 | 7
  RECIST v1.1 | 9.7 [3.7 to NA] — Not estimable. | NA — Not estimable. | 21.8 [5.8 to NA] — Not estimable. | 13.9 [3.8 to NA] — Not estimable.
  irRECIST | 13.0 [4.1 to NA] — Not estimable. | NA — Not estimable. | 22.1 [6.8 to NA] — Not estimable. | NA [4.6 to NA] — Not estimable.

21. Secondary Outcome: Time to Response (TTR) Based on RECIST Version 1.1 - Part 2
Description: TTR was the time to confirmed or unconfirmed complete response (CR) or partial response (PR) based on investigator assessment per RECIST v1.1 by tumor type. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must have decreased to normal size (short axis < 10 mm). All target lesions must have been assessed. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. All target lesions must have been assessed.
Time Frame: Baseline up to end of treatment in Part 2 (maximum of 851 days)
Population: as for outcome 5
Measure: Median (Full Range); unit: Months
Arm/Group | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 14 | 8
Months | 2.71 [1.4 to 12.0] | 2.33 [1.4 to 5.5]

22. Secondary Outcome: Time to Progression (TTP) Based on RECIST Version 1.1 and irRECIST - Part 2
Description: TTP was the time to objective progression. Objective progression was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum was observed during therapy), with a minimum absolute increase of 5 mm. TTP was analyzed by the Kaplan-Meier approach for each tumor type.
Time Frame: Baseline up to end of treatment in Part 2 (maximum of 851 days)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 67 | 38
Months
  RECIST v1.1 | 3.7 [1.9 to 5.7] | 3.7 [1.9 to 8.5]
  irRECIST | 6.5 [3.7 to 10.3] | 8.5 [2.5 to 19.4]

23. Secondary Outcome: Median Time to Death - Part 2
Description: Median time to death was analyzed by the Kaplan-Meier approach for each tumor type.
Time Frame: Baseline up to end of treatment in Part 2 (maximum of 851 days)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 68 | 39
Months | 14.7 [7.1 to NA] — Not estimable. | 10.9 [7.2 to 19.9]

24. Secondary Outcome: Probability of Survival at 6 Months, 1 Year, and 2 Years - Part 2
Description: Probability of survival was calculated from the product-limit method.
Time Frame: Baseline up to end of treatment in Part 2 (maximum of 851 days)
Population: Analysis population included all the randomized participants who received PF-06801591 and had at least 1 post-dose concentration measurement above the lower limit of quantification (LLQ).
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 68 | 39
Probability
  6 Months | 0.773 [0.647 to 0.859] | 0.711 [0.527 to 0.833]
  1 Year | 0.547 [0.407 to 0.667] | 0.471 [0.290 to 0.633]
  2 Years | 0.403 [0.265 to 0.537] | 0.286 [0.127 to 0.467]

25. Secondary Outcome: Trough PF-06801591 Concentrations (Ctrough) - Part 2
Description: Trough PF-06801591 Concentrations (Ctrough) - Part 2. Ctrough was directly observed from data.
Time Frame: Pre-dose on Day 1 of Cycles 2-6, 9, 12, 15, 18, 21, 24, and Follow-up Day 28 in Part 2
Population: Analysis population included all participants who received PF-06801591, had no protocol deviations affecting the pharmacokinetics (PK) assessment, and had at least 1 post-dose concentration measurement above lower limit of quantification.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC
Number analyzed (Participants) | 68 | 39
ug/mL
  Cycle 2 Day 1: number analyzed (Participants) | 58 | 35
  Cycle 2 Day 1 | 14.97 (48) | 14.34 (73)
  Cycle 3 Day 1: number analyzed (Participants) | 52 | 27
  Cycle 3 Day 1 | 22.54 (37) | 20.15 (84)
  Cycle 4 Day 1: number analyzed (Participants) | 42 | 18
  Cycle 4 Day 1 | 23.55 (53) | 23.77 (60)
  Cycle 5 Day 1: number analyzed (Participants) | 35 | 17
  Cycle 5 Day 1 | 23.58 (41) | 19.32 (186)
  Cycle 6 Day 1: number analyzed (Participants) | 29 | 13
  Cycle 6 Day 1 | 29.67 (36) | 17.13 (249)
  Cycle 9 Day 1: number analyzed (Participants) | 23 | 12
  Cycle 9 Day 1 | 29.01 (36) | 29.88 (30)
  Cycle 12 Day 1: number analyzed (Participants) | 18 | 8
  Cycle 12 Day 1 | 34.29 (16) | 12.74 (770)
  Cycle 15 Day 1: number analyzed (Participants) | 15 | 9
  Cycle 15 Day 1 | 40.90 (22) | 22.10 (56)
  Cycle 18 Day 1: number analyzed (Participants) | 12 | 6
  Cycle 18 Day 1 | 35.09 (25) | 20.17 (75)
  Cycle 21 Day 1: number analyzed (Participants) | 11 | 5
  Cycle 21 Day 1 | 27.16 (25) | 22.11 (55)
  Cycle 24 Day 1: number analyzed (Participants) | 7 | 3
  Cycle 24 Day 1 | 30.81 (16) | 38.02 (38)
  Follow-up Day 28: number analyzed (Participants) | 5 | 3
  Follow-up Day 28 | 43.62 (33) | 35.17 (32)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug (up to a maximum of 237 weeks).
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Groups:
- Part 1: PF-06801591 IV Total: Participants received PF-06801591 IV every 3 weeks for 21-day cycles in Part 1. (up to a maximum of of 233 weeks)
- Part 1: PF-06801591 IV and SC Total: Participants received PF-06801591 IV every 3 weeks for 21-day cycles or SC every 4 weeks for 28-day cycles in Part 1. (up to a maximum of 233 weeks)
- Part 2: PF-06801591 NSCLC and UC Total: Participants with NSCLC or UC received PF-06801591 300 mg SC every 4 weeks for 28-day cycles in Part 2. (up to a maximum of 126 weeks)
Arm/Group | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) | Part 1: PF-06801591 1 mg/kg (IV) | Part 1: PF-06801591 3 mg/kg (IV) | Part 1: PF-06801591 10 mg/kg (IV) | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) | Part 1: PF-06801591 IV Total | Part 1: PF-06801591 IV and SC Total | Part 2: PF-06801591 300 mg (SC) for NSCLC | Part 2: PF-06801591 300 mg (SC) for UC | Part 2: PF-06801591 NSCLC and UC Total
All-Cause Mortality (participants affected / at risk) | 1/2 | 6/8 | 5/8 | 6/7 | 10/15 | 18/25 | 28/40 | 33/68 | 21/38 | 54/106
Serious Adverse Events (participants affected / at risk) | 1/2 | 3/8 | 3/8 | 3/7 | 3/15 | 10/25 | 13/40 | 18/68 | 13/38 | 31/106
Other Adverse Events (participants affected / at risk) | 2/2 | 7/8 | 8/8 | 7/7 | 15/15 | 24/25 | 39/40 | 59/68 | 33/38 | 92/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) (N=2) | Part 1: PF-06801591 1 mg/kg (IV) (N=8) | Part 1: PF-06801591 3 mg/kg (IV) (N=8) | Part 1: PF-06801591 10 mg/kg (IV) (N=7) | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) (N=15) | Part 1: PF-06801591 IV Total (N=25) | Part 1: PF-06801591 IV and SC Total (N=40) | Part 2: PF-06801591 300 mg (SC) for NSCLC (N=68) | Part 2: PF-06801591 300 mg (SC) for UC (N=38) | Part 2: PF-06801591 NSCLC and UC Total (N=106)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 1 | 2 | 0 | 4 | 4 | 3 | 2 | 5
Mucosal ulceration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: PF-06801591 0.5 mg/kg (Intravenously [IV]) (N=2) | Part 1: PF-06801591 1 mg/kg (IV) (N=8) | Part 1: PF-06801591 3 mg/kg (IV) (N=8) | Part 1: PF-06801591 10 mg/kg (IV) (N=7) | Part 1: PF-06801591 300 mg (Subcutaneously [SC]) (N=15) | Part 1: PF-06801591 IV Total (N=25) | Part 1: PF-06801591 IV and SC Total (N=40) | Part 2: PF-06801591 300 mg (SC) for NSCLC (N=68) | Part 2: PF-06801591 300 mg (SC) for UC (N=38) | Part 2: PF-06801591 NSCLC and UC Total (N=106)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 3
Bundle branch block (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 8 | 3 | 11
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0 | 1 | 1 | 3 | 4 | 5 | 4 | 9
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Punctate keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 1 | 4 | 5 | 1 | 2 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 4 | 2 | 3 | 2 | 11 | 13 | 2 | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 3 | 2 | 4 | 8 | 12 | 4 | 5 | 9
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 2 | 4 | 1 | 1 | 2
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 3 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 0 | 6 | 6 | 12 | 5 | 3 | 8
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 3 | 4 | 0 | 0 | 0
Pancreatic failure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 5 | 7 | 12 | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 7 | 6 | 13
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 0 | 4
Chills (General disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 3 | 8 | 3 | 11
Generalised oedema (General disorders) | 2 | 3 | 4 | 4 | 5 | 13 | 18 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 3
Injection site pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 1 | 0 | 1 | 1 | 4 | 5 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Oedema (General disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 3 | 2 | 5
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 8 | 3 | 11
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 1 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1 | 3 | 3 | 6 | 2 | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 1 | 2 | 4 | 6 | 2 | 5 | 7
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1 | 2 | 3 | 2 | 2 | 4
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 8 | 2 | 10
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 6 | 4 | 10
Aspartate aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 2 | 1 | 4 | 5 | 7 | 2 | 9
Blood albumin decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Blood alkaline phosphatase abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 5 | 2 | 7
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 5 | 0 | 5
Blood creatinine increased (Investigations) | 2 | 1 | 1 | 0 | 2 | 4 | 6 | 3 | 3 | 6
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 2
Blood magnesium increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 3 | 0 | 1 | 3 | 4 | 0 | 1 | 1
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 6
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 5 | 4 | 9
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 4
Weight decreased (Investigations) | 1 | 0 | 1 | 1 | 2 | 3 | 5 | 4 | 2 | 6
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 1 | 0 | 7 | 6 | 13 | 9 | 3 | 12
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 3 | 4 | 7 | 2 | 1 | 3
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 3 | 3 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 1 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 3 | 3 | 6 | 1 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 0 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1 | 2 | 6 | 8 | 4 | 4 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 4 | 4 | 8 | 3 | 6 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 2 | 2 | 4
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 1 | 0 | 5 | 5 | 3 | 1 | 4
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 3 | 4 | 3 | 2 | 5
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 2 | 0 | 0 | 3 | 3 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 2
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0 | 0 | 3 | 3 | 6 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 1 | 1 | 3 | 4 | 6 | 0 | 6
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 2
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 4
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 0 | 3 | 3 | 1 | 1 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 4 | 2 | 6
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1 | 4 | 6 | 10 | 6 | 2 | 8
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2 | 5 | 6 | 11 | 10 | 0 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 3 | 4 | 1 | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 5
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 7 | 1 | 8
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 4 | 4 | 8 | 4 | 12
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 5 | 2 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 3
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 3
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Peripheral embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Shock (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 12 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT02573259/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT02573259/SAP_001.pdf